CLINICAL TRIAL: NCT01174797
Title: Evaluation of Microvolt T-Wave Alternans Testing for the Detection of Active Ischemia in Patients With Known or Suspected Coronary Artery Disease: A Feasibility Study
Brief Title: Evaluation of Microvolt T-Wave Alternans(MTWA) Testing for the Detection of Active Ischemia
Acronym: MTWA-CAD
Status: Completed | Type: Observational
Sponsor: Cambridge Heart Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 60-0001-001
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients being evaluated for active ischemia: Subjects with known or suspected CAD who are scheduled to undergo routine exercise MPI or stress echocardiography for the detection of active ischemia are eligible for enrollment.

SUMMARY:
MTWA-CAD is a feasibility study designed to evaluate Microvolt T-Wave Alternans (MTWA) testing for the purpose of detecting active ischemia in patients with known or suspected coronary artery disease (CAD). MTWA is a subtle, alternating pattern in the T wave portion of the surface electrocardiogram (ECG) that is associated with increased risk of ventricular tachyarrhythmias and sudden cardiac arrest (SCA).

DETAILED DESCRIPTION:
Ischemia, a common trigger for arrhythmias, is a well-documented cause of repolarization alternans. Human studies have shown that active ischemia can be associated with visible as well as microvolt-level T-wave alternans. While MTWA testing is traditionally used to evaluate arrhythmic risk, this known association with ischemia may allow MTWA testing to be used as a diagnostic tool to detect underlying CAD. The MTWA-CAD study will assess the feasibility of this concept by measuring MTWA during routine nuclear stress testing or stress echocardiography with treadmill exercise. This is a feasibility study designed to verify preliminary observations under controlled environments and to generate hypotheses, endpoints, and sample sizes for future investigations.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above, or of legal age to give informed consent specific to state and national law
* Willing and capable of providing informed consent
* Willing and capable of undergoing a SPECT MPI exercise test (or stress echo) at an approved clinical investigational center
* In normal sinus rhythm at the time of the exercise test
* A life expectancy of more than 6 months

Exclusion Criteria:

* In atrial fibrillation at the time of the exercise test
* Left bundle branch block (precludes ST segment measurement)
* Pacemaker-dependent
* Life expectancy of less than 6 months
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with known or suspected CAD who are scheduled to undergo routine exercise MPI or stress echocardiography testing for the detection of active ischemia in a cardiology practice or hospital setting.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2010-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward J Kosinski, MD, Principal Investigator — Connecticut Clinical Research, LLC
Locations (2):
- United States (2):
  - Connecticut Clinical Research, LLC, Bridgeport, Connecticut
  - Northwest Houston Heart Center, Tomball, Texas